CLINICAL TRIAL: NCT00005038
Title: A Randomized Phase II Study to Evaluate the Efficacy of Combined Immunotherapy With Subcutaneous Interleukin-2 and Maxamine in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Interleukin-2 With or Without Histamine Dihydrochloride in Treating Patients With Metastatic Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067627; CHNT-IL2-MAXAMINE; EU-99048; MAXIM-MP-502
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-06

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Histamine

INTERVENTIONS:
Biological: aldesleukin
Drug: histamine dihydrochloride

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill kidney cancer cells. Histamine dihydrochloride may prolong survival and improve quality of life in patients with metastatic kidney cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of interleukin-2 with or without histamine dihydrochloride in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical efficacy and safety of subcutaneous (SC) histamine dihydrochloride given in conjunction with SC recombinant human interleukin-2 in patients with stage IV renal cell carcinoma in terms of survival at 1 year, objective tumor response rate, duration of response, and median survival.

OUTLINE: This is a randomized, open label study. Patients are randomized to receive interleukin-2 (IL-2) with or without histamine dihydrochloride.

* Arm I: Patients receive IL-2 subcutaneously (SC) once daily and histamine dihydrochloride SC twice daily on days 1-5 of weeks 1-3 followed by 2 weeks of rest.
* Arm II: Patients receive IL-2 as in arm I. Treatment continues for a minimum of 2 courses in both arms in the absence of unacceptable toxicity or disease progression.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 60 patients (30 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic renal cell carcinoma
* Bidimensionally measurable disease
* No clinical evidence of CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Hemoglobin greater than 10.0 g/dL
* WBC greater than 3,000/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* PTT normal
* Bilirubin less than 1.25 times upper limit of normal (ULN)

Renal:

* Creatinine less than 1.5 times ULN

Cardiovascular:

* No abnormal cardiac function by resting ECG

Pulmonary:

* FEV and FVC at least 70% predicted
* SaO2 at least 90% by pulse oximetry

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No clinically significant acute viral, bacterial, or fungal infection requiring specific therapy
* No pheochromocytoma
* No glaucoma
* No other concurrent ongoing active malignancy except carcinoma in situ of the cervix or localized squamous or basal cell carcinoma of the skin
* No serious recent nonmalignant medical complication that would preclude study therapy
* No organ grafts except skin grafts, blood transfusions, or bone marrow or stem cell transplantation
* No prior documented asthma or systemic allergic reaction within past 5 years
* No history of seizures, CNS disorders, or psychiatric disability that would preclude study compliance
* No medical, sociologic, or psychological impediment that would preclude study compliance
* No active peptic or esophageal ulcer disease
* No prior peptic or esophageal ulcer disease with history of bleeding
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin)
* No concurrent chemotherapy

Endocrine therapy:

* At least 24 hours since prior steroids
* No concurrent steroids including steroid therapy for documented adrenal failure or septic shock
* Concurrent noncorticosteroid hormones for nonmalignancy conditions allowed

Radiotherapy:

* At least 4 weeks since prior extensive radiotherapy
* No concurrent radiotherapy to measurable malignant masses

Surgery:

* Not specified

Other:

* At least 24 hours since prior beta blockers or clonidine
* No other concurrent systemic antimalignancy therapy
* No other concurrent antitumor agents
* No other concurrent investigational agents
* No concurrent beta blockers or clonidine
* No concurrent H2 receptor antagonists (e.g., Zantac, Tagamet) (arm I only)
* No concurrent antihistamines except to treat acute colds or allergy symptoms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Middleton, MD, PhD, MBChB, MRCP, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital N.H.S. Trust, Manchester, England, United Kingdom